CLINICAL TRIAL: NCT03468413
Title: A Randomised, First-in-human, Double-blinded, Placebo-controlled Study to Determine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of CP1050 in Healthy Subjects; Including the Effect of Food and Gender on the Pharmacokinetics and Pharmacodynamics of a Single Dose of CP1050 in Healthy Subjects
Brief Title: A First-in-human Phase 1 Study of CP1050
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Curadim Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP1050-E101
Record Dates: First submitted 2018-02-22; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Healthy Subjects
Keywords: CP1050; Phase 1; Healthy subjects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single ascending dose, CP1050 or Placebo (Experimental)
  Interventions: Drug: CP1050 or Placebo
- Multiple ascending dose, CP1050 or Placebo (Experimental)
  Interventions: Drug: CP1050 or Placebo

INTERVENTIONS:
Drug: CP1050 or Placebo — Randomised, double-blinded, placebo-controlled

SUMMARY:
This is a Phase I, first-in-human, double-blind, single-centre, randomised, placebo-controlled, single and multiple oral dose study in healthy subjects conducted in 4 parts (Part 1; Single-ascending dose, Part 2; Food-effect evaluation, Part 3; Gender-effect evaluation, Part 4; Multiple-ascending dose).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian males or females between 18 and 55 years of age (inclusive).
* A body weight of ≥60 kg for males and ≥50 kg for females, with a body mass index (BMI) ranging from 18.0 to 30.0 kg/m2 (inclusive).
* Healthy and free from clinically significant illness or disease.

Exclusion Criteria:

* Presence or history of any clinically significant disease that could interfere with the objectives of the study or the safety of the subject in the opinion of the Investigator.
* Participation in more than 3 clinical studies involving administration of an IMP in the past one year, or any study within 12 weeks.
* Clinically significant abnormalities in ECG or laboratory tests.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 116 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of any drug-related adverse events | Up to 21 days
  To evaluate the safety and tolerability of CP1050 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of adverse events
Number of subjects with abnormal vital signs (systolic and diastolic blood pressure, pulse rate, respiratory rate and oral body temperature) | Up to 21 days
  To evaluate the safety and tolerability of CP1050 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of vital signs
Number of subjects with abnormal clinical laboratory tests (including clinical chemistry, haematology and urinalysis) | Up to 21 days
  To evaluate the safety and tolerability of CP1050 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of clinical laboratory tests
Number of subjects with abnormal 12-lead safety ECG (including heart rate, RR interval, PR interval, QRS duration, QT interval, and QT interval corrected for heart rate using Fridericia's method [QTcF]) | Up to 21 days
  To evaluate the safety and tolerability of CP1050 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of 12-lead safety ECG
Number of subjects with abnormal 12-lead continuous (24-hour) ECG (including mean hourly heart rate and incidence of arrhythmia assessed as per the ECG Alert Criteria) | Up to 21 days
  To evaluate the safety and tolerability of CP1050 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of 12-lead continuous (24-hour) ECG
Number of subjects with abnormal Pulmonary function tests (including FEV1, FVC, FEF25-75 and DLCO [Part 4 only]) | Up to 21 days
  To evaluate the safety and tolerability of CP1050 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of pulmonary function tests
Number of subjects with abnormal ophthalmological findings assessed by fundoscopy or OCT | Up to 21 days
  To evaluate the safety and tolerability of CP1050 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of ophthalmological assessments
Number of subjects with abnormal physical examinations | Up to 21 days
  To evaluate the safety and tolerability of CP1050 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of physical examinations

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 21 days
Area under the plasma concentration-time curve (AUC) | Up to 21 days
Time of maximum observed plasma concentration (Tmax) | Up to 21 days
Apparent plasma terminal elimination half-life (T1/2) | Up to 21 days
The lowest absolute value of lymphocytes at postdose (nadir) | Up to 21 days
The lowest percentage of baseline (nadir [%]) | Up to 21 days
Time of nadir (Tnadir) | Up to 21 days
Area under the effectiveness curve (AUCE) | Up to 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit (CRU) Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No